CLINICAL TRIAL: NCT04093726
Title: Effect of Chewing Lollipop on Gastric Residual Volume
Brief Title: Lollipop on Gastric Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: XJH-A-20190916-2
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Gastric Volume

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lollipop (Experimental)
  Interventions: Other: lollipop
- control (No Intervention)

INTERVENTIONS:
Other: lollipop — chewing lollipop for 20min
  Arms: lollipop

SUMMARY:
To observe the effect of chewing lollipop on residual gastric volume in healthy volunteers with fasting.

ELIGIBILITY:
Inclusion Criteria:

* volunteer aged 18 years-45 years old
* volunteer with a body mass index between 18 and 28 kg/m2

Exclusion Criteria:

* those with history of diabetes mellitus
* those with gastric diseases
* those with history of gastro-intestinal surgery
* those with history of smoking
* those with use of gastric mobility medicines
* those with pregnancy or breeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2019-12-22 (Actual); Study Completion 2019-12-22 (Actual)

PRIMARY OUTCOMES:
residual gastric volume at 30 minutes after chewing lollipop | from starting chewing lollipop to 30 minutes after chewing, on an average of 30 minutes

SECONDARY OUTCOMES:
residual gastric volume at 2 hours after chewing lollipop | from starting chewing lollipop to 2 hours after chewing, on an average of 2 hours
residual gastric volume at 1 hour after chewing lollipop | residual gastric volume at 1 hour after chewing lollipop
time to peak gastric volume | from starting chewing lollipop to gastric volume reaching peak , on an average of 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided
Data of primary and secondary outcomes could be shared

REFERENCES:
- [Result] Schoenfelder RC, Ponnamma CM, Freyle D, Wang SM, Kain ZN. Residual gastric fluid volume and chewing gum before surgery. Anesth Analg. 2006 Feb;102(2):415-7. doi: 10.1213/01.ane.0000189218.07293.6e. PMID 16428535